CLINICAL TRIAL: NCT02844894
Title: The Effects of Preintubation Esmolol and and Dexmedotimidine on Ischmeia Modified Albumin Levels
Brief Title: Hemodynamic Response to Intubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Perihan Ekmekçi, Associate Professor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RespToIntubation
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Intubation
Keywords: intubation, ischemia modified albumine, dexmedetomidine, esmolol
MeSH Terms: interventions — Dexmedetomidine; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- dexmedetomidine (Experimental): 0.5 mcg/kg dexmedetomidine in 20 ml normal saline will be infused in 5 minutes before intubation
  Interventions: Drug: Dexmedetomidine
- Esmolol (Experimental): 0.5 mg/kg esmolol in 20 ml normal saline will be infused in 5 minutes before intubation
  Interventions: Drug: Esmolol
- Placebo (Placebo Comparator): 20 ml normal saline infused in 5 minutes before intubation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: dexmedetomidine
Drug: Esmolol
  Arms: Esmolol
Drug: Placebo — normal saline
  Arms: Placebo

SUMMARY:
This study investigates the effects of dexmedetomidine and esmolol given intravenously before intubation on sympathetic response caused by intubation itself. Half the patients will recevice dexmedetomidine and the other half will receive dexmedetomidine. Ischemia modified albumine levels will be measured

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery under general anesthesia

Exclusion Criteria:

* Patient refusal
* Morbid obesity (BMI>30)
* Advanced systemic disease
* Hypoalbumiemia
* beta-blocker usage
* Anticipated difficult ventilation and/or intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
ischemia modified albumine | 10 minutes after endotracheal intubation
  ischemia modified albumine levels will be measured as a response to intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yallapragada SV, Vidadala KS, Vemuri NN, Shaik MS. Comparison of the efficacy of dexmedetomidine with that of esmolol in attenuating laryngoscopic and intubation response after rapid sequence induction. Anesth Essays Res. 2014 Sep-Dec;8(3):383-7. doi: 10.4103/0259-1162.143154. PMID 25886340